CLINICAL TRIAL: NCT06516419
Title: Development of Products Based on Secretom From Stem Cell Conditioned Medium for Melasma Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr.dr.Irma Bernadette, SpKK (K) (Other)
Responsible Party: Sponsor-Investigator, Dr.dr.Irma Bernadette, SpKK (K), Prof. Dr. dr. Irma Bernadette S. Sitohang, SpKK(K), Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Secretome
Record Dates: First submitted 2024-07-08; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Secretom group) (Experimental): Group A, the treatment group, used Secretom 2ml Intradermal injection, Sunscreen in the morning and used Tretinoin cream 0,05% at night and cleanser which was used in the morning and evening before using the cream.
  Interventions: Drug: Concentrated secretome Injection 2mL
- Group B (Triple Combination Group) (Experimental): Group B, the treatment group, getting sunscreen cream in the morning and triple combination (Refaquin) cream at night and facial soap that can be used in the morning and evening.
  Interventions: Drug: Triple Combination Cream
- Group C (Tranexamic Acid Group) (Experimental): Group C, the treatment group, used Intradermal Injection of Tranexamic Acid 10mg/mL and 25mg/mL split face , Sunscreen in the morning and used Tretinoin cream 0,05% at night and cleanser which was used in the morning and evening before using the cream.
  Interventions: Drug: Tranexamic acid injection

INTERVENTIONS:
Drug: Concentrated secretome Injection 2mL — The secretome used in this research comes from mesenchymal stem cells from adipose tissue produced by IPT RSCM Stem Cell Medical Technology. The secretome produced by mesenchymal stem cells is collected, centrifuged to separate it from debris, and followed by filtration with a 0.22 μm pore filter to ensure sterility. Next, the concentration process is carried out using tangential flow filtration with the Spin-X UF 500® concentrator, packaged, and stored at -80 degrees Celsius. The product used is a sterile product, which is tested for sterility and total protein content. When it is to be used, the secretome is removed from the freezer, warmed (thawing), and injected into the patient according to a predetermined method.
  Arms: Group A (Secretom group)
Drug: Tranexamic acid injection — 1. Tranexamic acid 25 mg/ml is prepared by taking tranexamic acid in a vial 250 mg/5 ml as much as 0.5 ml (25 mg) using a 1 ml syringe and diluted with 0.5 ml 0.9% NaCl solution just before being injected into the SP.
  2. Tranexamic acid 10 mg/ml is prepared by taking 0.2 ml (10 mg) of AT in a 250 mg/5 ml vial using a 1 ml syringe and diluting it with 0.8 ml of 0.9% NaCl solution for a moment. before injection into the Subject
  2. Tranexamic acid 10 mg/ml is prepared by taking 0.2 ml (10 mg) of AT in a 250 mg/5 ml vial using a 1 ml syringe and diluting it with 0.9% normal saline (NS) 0.8 ml just before injection into the Subject
  Arms: Group C (Tranexamic Acid Group)
Drug: Triple Combination Cream — 1. Apply sunscreen SPF ≥30 in the morning on 2 knuckles
  2. Apply triple combination cream (Refaquin) containing hydroquinone 40 mg, tretinoin 0.5 mg, and fluocinolone acetonide 0.1 mg at night all over the face except the area around the eyes, 1 fingertip unit (FTU) or 1 knuckle.
  Arms: Group B (Triple Combination Group)

SUMMARY:
This research is a clinical study with a single-blind randomized clinical trial design (randomized controlled trial) in RSCM-FKUI

This study aims to Assess the effectiveness and safety of intradermal concentrated secretome injection therapy, triple combination cream, and intradermal tranexamic acid injection in melasma patients, determine the quality of life profile of melasma patients after triple combination cream therapy in melasma therapy, and determine SOD levels in melasma patients.

This research will be attended by 90 research subjects

DETAILED DESCRIPTION:
Melasma is a pigmentation disorder in the form of brownish macules with irregular edges caused by dysfunction of melanogenesis. Melasma occurs more often in women with Fitzpatrick skin types IV-VI, namely those of Asian, Hispanic and African descent, especially on parts of the face that are exposed to sunlight.

The therapeutic modality that is being developed for melasma therapy is the secretome. The secretome is a bioactive molecule secreted by Mesenchymal Stem Cells in a conditioned medium containing a large number of growth factors, cytokines, and various macromolecules, and extracellular vesicles including microvesicles and exosomes that can stimulate various biological reactions, especially in modulating various new tissue formations.

So far there have been no clinical trial studies comparing the application methods of intradermal concentrated secretome injection, triple combination cream, and intradermal tranexamic acid injection as melasma therapy in Indonesia and the quality of life profile of melasma patients tested using the MELASQoL-INA questionnaire is not yet known.

This research is a study using a Randomized Controlled Trial (RCT) design that compares intradermal concentrated secretome injection, triple combination cream, and intradermal injection of tranexamic acid.

This study was single-blind randomized to investigators. The secretome of mesenchymal stem cells from adipose tissue will be produced by IPT Stem Cell Medical Technology RSCM-FKUI, CMU 2 Building, 5th Floor, while research on subjects with melasma will be carried out at the RSCM Dermatology and Venereology Polyclinic

Research subjects were randomized to determine the group for intradermal concentrated secretome injection, triple combination cream, and intradermal tranexamic acid injection.

Subjects will be divided into 30 people per group.

The research evaluation time is 12 weeks. The secretome injection group (A) and the tranexamic acid injection group (C) will be given 0.5% Tretinoin cream for 2 weeks as preparation.

Next, all SP groups A, B, and C will undergo an initial physical examination in the form of a physical examination, clinical photos, mMASI score, MelasQOL-INA, dermoscopy, Wood's lamp, and mexameter.

Group A evaluation will be carried out every 4 weeks, namely weeks 0, 4, 8, 12 with Secretome injections 3 times, namely at weeks 0, 4 and 8. Subjects are given facial wash, sunscreen and 0.5% tretinoin cream at night. day

Group B evaluation will be carried out every 4 weeks, namely weeks 0, 4, 8, 12. Subjects were given facial wash, sunscreen, and Refaquin cream (triple combination) for the night

Group C evaluation will be carried out every 2 weeks, namely weeks 0, 2, 4, 6, 8, and 12. Subjects are given facial wash, sunscreen, and 0.5% tretinoin cream at night.

Each evaluation will be checked:

* Physical examination
* mMASI score
* PtGA
* mexameter examination

Data is recorded in research status which is then compiled into a master table. The research results are attached in the form of narratives, tables and graphs. Data were processed statistically using STATA v.16 (StataCorpTM, USA).

The characteristics of the research subjects are presented in the characteristics table. Characteristics with categorical data are presented in the form of frequencies and percentages. Numerical data was subjected to normality analysis using the Kolmogorov Smirnov test and for numerical data with a normal distribution it was presented in the form of mean and standard deviation, while for non-normal distribution it was presented in the median and minimum and maximum values.

Comparison of mMASI scores, melanin index, erythema index, speed of decline between the three research groups, was analyzed using the unpaired t test. Data that is not normally distributed uses an alternative test, namely the Mann Whitney test. Comparison of mMASI scores, melanin index, and erythema index at each examination time with baseline were analyzed using the paired t test. Data that is not normally distributed uses an alternative test, namely the Wilcoxon test. Comparison of the proportion of telangiectasis scores between the intervention and control groups was analyzed using the Chi-square test.

The Pearson test is used to assess the correlation between mMASI and MELASQoL-INA scores if a normal data distribution is obtained, while the Spearman test is used if the data distribution is not normal. The test results obtained are in the form of a correlation coefficient (r) which is in the range -1 and 1. The r value which is in the range 0.1-0.3 indicates the correlation between the two variables is weak, the range 0.4-0.6 indicates a moderate correlation , a range of 0.6-0.9 indicates a strong correlation, and 1 indicates a perfect correlation. The value of statistical significance in the research is determined

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with melasma.
* Women without melasma and have areas of skin that are clinically free of lesions for SP control.
* 30-60 years old.
* Fitzpatrick skin type IV-V.
* Willing to be a research subject by signing a research consent form (Informed Consent).

Exclusion Criteria:

* Pregnant and breastfeeding women.
* Currently using hormonal contraception or have ever used contraception hormones in the last 6 months.
* Using topical therapy for melasma, for example corticosteroids, tretinoin, hydroquinone, and other therapies that whiten or brighten the skin in the last 2 weeks.
* Using topical triple combination cream therapy for at least 3 months and did not show significant improvement
* Using systemic therapy for melasma, for example antioxidants or tranexamic acid in the last 4 weeks.
* History of superficial peeling therapy in the last 4 weeks.
* History of deep peeling therapy, laser or mechanical abrasion in the last 6 months.
* Using drugs that are photosensitizers such as tetracycline, phenytoin, carbamazepine, spironolactone.
* History of blood clotting disorders or on blood thinning therapy.
* Allergy to tranexamic acid.
* Have other skin complaints that may interfere with the evaluation of melasma, for example post-inflammatory hyperpigmentation, Hori's nevus, Ota's nevus, pigmented contact dermatitis, and other pigmentation disorders
* Difficulty complying with treatment.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Change of Melasma Severity based on modified Melasma Severity Index (mMASI) score. | re-evaluation on day 14, 28, 42, 56 and day 84 of therapy
  The range of values for mMASI is between 0 and 24 which can then be divided into mild melasma (0-8), moderate (8-16), and severe (16-24).
  improvement occurs if the mMASI score decreases by <50% from the previous visit worsening if score persists or mMASI Score Increase >50%
Change of Melasma Severity based on Patient's Tolerability Assesment (PtGA). | re-evaluation on day 14, 28, 42, 56 and day 84 of therapy
  one method of evaluating the response to therapy in melasma which is assessed subjectively by the patient. The response to therapy can be assessed as follows
  No or slight response: < 25% improvement Moderate response: 25% - 50% improvement Good response: 50% improvement - < 75% Excellent response: improvement > 75% The response is said to be good if the score is above 50% since the previous visit
Change of Melasma Severity based on Dermoscopy | re-evaluation on day 84 of therapy
  based on Dermoscopy
  Telangiectasis score assessment using a 5-point dermoscopy-scale:
  0 = No visible capillaries.
  1 = Elongated capillaries accompanied by dilation, not visible to the naked eye. 2 = Moderate telangiectasis that is beginning to be visible to the naked eye.
  3 = Severe telangiectasis characterized by reduced capillary loops. 4 = Very severe telangiectasis characterized by dilatation and loss of capillary loops.
Change of Melasma Severity based on Wood's Lamp | re-evaluation on day 84 of therapy
  Epidermal Type/ Dermal Typed/ Mixed Typed
Compare Quality Of Life based on MelasQoL Score | re-evaluation on day 84 of therapy
  based on MelasQoL Score minimum score: 7 maximum score : 70
Change of Melanin Index Based on Mexameter | re-evaluation on day 14, 28, 42, 56 and day 84 of therapy
  improves if there is a decrease in melanin levels > 50% from the initial visit It is said to be bad or persistent if there is no decrease in melanin levels or there is a decrease of <50%
Change of Erytema Index Based on Mexameter | re-evaluation on day 14, 28, 42, 56 and day 84 of therapy
  improves if there is a decrease in Erytema levels > 50% from the initial visit It is said to be bad or persistent if there is no decrease in erythema levels or there is a decrease of <50%

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - Clinical Research Supporting Unit- Faculty of Medicine, University of Indonesia, Jakarta Pusat, DKI Jakarta
  - Dr. Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta

IPD SHARING:
Plan to Share IPD: Undecided